CLINICAL TRIAL: NCT02028897
Title: Comparison of Alternative Embryo Culture Systems
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce Shapiro M.D. (Industry)
Responsible Party: Sponsor-Investigator, Bruce Shapiro M.D., Medical Director, Fertility Center of Las Vegas
Organization: Fertility Center of Las Vegas (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAIRB-13-0040
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
Keywords: In vitro fertilization; IVF; Embryo culture; Blastocyst transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional embryo culture (Active Comparator): Conventional embryo culture in dishes, in droplets under oil.
  Interventions: Other: Conventional embryo culture
- Alternative embryo culture (Experimental): Embryo culture in system using small enclosed containers
  Interventions: Other: Enclosed embryo culture

INTERVENTIONS:
Other: Conventional embryo culture
  Arms: Conventional embryo culture
Other: Enclosed embryo culture
  Arms: Alternative embryo culture

SUMMARY:
This study will compare two alternative embryo culture systems. Embryos from each patient will be randomly assigned to one of two systems. One group will be cultured conventionally in oil-covered droplets in dishes. The other group will be assigned to an enclosed system.

DETAILED DESCRIPTION:
Qualifying and consenting IVF patients will have approximately half of their developing embryos cultured in droplets covered with oil. The other approximate half of their embryos will be cultured in small enclosed containers. Embryo assignments will be at random. Regardless of culture system, all embryos will be cultured from the bipronuclear stage to the blastocyst stage in the same (Global) media, without the usual refreshing of media on day 3.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 to 40, seeking IVF treatment
* Ability to understand English (to obtain informed consent)
* Use of an oocyte donor, sperm donor, gestational carrier, and/or genetic testing (with blastocyst biopsy only) are allowed.

Exclusion Criteria:

* Diminished ovarian reserve as evidenced by either elevated cycle day 3 follicle stimulating hormone (FSH) level (≥10 IU/L) or low antral follicle count (<8 antral follicles)
* Fewer than five (5) bipronuclear oocytes
* Day 3 embryo biopsy for any reason
* No minors may enroll

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Blastulation rate | 5 days (sixth day of embryo development)
  Proportion of cultured embryos that form blastocysts.

SECONDARY OUTCOMES:
Blastocyst morphology | 5 days (sixth day of development)
  Inner cell mass size, number of trophectoderm cells, blastocyst diameter
IVF outcome | 7 weeks post-transfer
  The result of the IVF cycle as no pregnancy, early pregnancy loss, or ongoing pregnancy at 10 weeks gestation (about 7 weeks post-transfer).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shapiro, MD, PhD, Principal Investigator — Fertility Center of Las Vegas
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States